CLINICAL TRIAL: NCT03871387
Title: The Effects of Deep Neuromuscular Blockade During Robot-assisted Transaxillary Thyroidectomy on Postoperative Pain and Sensory Change; Prospective Randomized Control Trial
Brief Title: The Effects of Deep Neuromuscular Blockade During Robot-assisted Transaxillary Thyroidectomy on Postoperative Pain and Sensory Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2018-0963
Record Dates: First submitted 2019-02-26; First posted 2019-03-12 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Thyroid Neoplasms
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: 1. Deep group
     * Continuous rocuronium infusion during surgery
     * Maintain TOF = 0 & PTC= 1~2 (Deep neuromuscular block)
  2. Control group
     * Continuous rocuronium infusion during surgery
     * Maintain TOF 1~2 (Moderate neuromuscular block)
Who Masked: Participant, Care Provider
Masking Description: Participants and Care Providers will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep Block Group (Experimental): * Continuous Rocuronium infusion during surgery
  * Maintain TOF = 0 & PTC= 1~2
  * At the end of surgery, IV Sugammadex injection to reverse muscle relaxation. (Sugammadex dose = 2mg/kg at TOF ≥2 or 4mg/kg at TOF < 2)
  Interventions: Drug: Deep Group
- Moderate Block Group (Active Comparator): * Continuous Rocuronium infusion during surgery
  * Maintain TOF 1~2
  * At the end of surgery, IV Sugammadex injection to reverse muscle relaxation. (Sugammadex dose = 2mg/kg at TOF ≥2 or 4mg/kg at TOF < 2)
  Interventions: Drug: Control Group

INTERVENTIONS:
Drug: Deep Group — * Continuous Rocuronium (Rocnium®, Hanlim Pharm. Co., Ltd., South Korea) infusion during surgery
  * Titrate Rocuronium (Rocnium®) infusion rate to maintain TOF = 0 & PTC= 1~2 (TOF = train-of-four. PTC = post-tetanic count)
  * TOF and PTC are assessed by acceleromyography (TOF-Watch® SX, Organon Ltd., Drynam Road, Swords, Co. Dublin, Ireland).
  * At the end of surgery, IV Sugammadex (Bridion®, Merck Sharp and Dohme [MSD], Oss, the Netherlands) injection to reverse muscle relaxation.
  * Sugammadex dose = 2mg/kg at TOF ≥2 or 4mg/kg at TOF < 2
  Other Names: Deep Neuromuscular Block
  Arms: Deep Block Group
Drug: Control Group — * Continuous Rocuronium (Rocnium®, Hanlim Pharm. Co., Ltd., South Korea) infusion during surgery
  * Titrate Rocuronium (Rocnium®) infusion rate to maintain TOF = 1~2
  * TOF and PTC are assessed by acceleromyograph (TOF-Watch® SX, Organon Ltd., Drynam Road, Swords, Co. Dublin, Ireland).
  * At the end of surgery, IV Sugammadex (Bridion®, Merck Sharp and Dohme [MSD], Oss, the Netherlands) injection to reverse muscle relaxation.
  * Sugammadex dose = 2mg/kg at TOF ≥2 or 4mg/kg at TOF < 2
  Other Names: Moderate Neuromuscular Block
  Arms: Moderate Block Group

SUMMARY:
As robotic surgery has been applied to various surgeries, the minimally invasive surgery is rapidly evolving. In particular, robot-assisted thyroidectomy is one of the leading techniques in minimally invasive surgery fields. Robot-assisted transaxillary thyroidectomy dramatically improves the cosmetic satisfaction, showing no difference in cancer control and safety comparing with conventional open thyroidectomy. However, some studies have shown that many patients complained of chest pain after robot-assisted thyroidectomy, and about 20% of patients suffered chronic pain even after three months of surgery. This might be due to the flap formation during robot-assisted thyroidectomy.

Robot-assisted transaxillary thyroidectomy does not provide visibility by injecting CO2. But it provides visibility using Chung's retractor system to make a flap between the pectoralis major muscle and subcutaneous fat layer. The flap is formed from the incision of axilla to the anterior neck to approach the thyroid gland. In this progress, it requires considerable force to maintain the Chung's retractor system, and additional pressure may be applied to the subcutaneous fat and skin constituting the skin flap. The pressure applied to the skin flap may be associated with postoperative pain and sensory abnormality, but it has not been studied yet.

Deep neuromuscular blockade The neuromuscular block for muscle relaxation during surgery is essential for general anesthesia. In general, a neuromuscular block agent is used to induce intubation during induction of anesthesia. Continuous or single injection of neuromuscular block agent is then carried out as needed during the operation.

The effect of deep neuromuscular blockade on laparoscopic surgery using carbon dioxide has already been studied. Deep neuromuscular blockade on laparoscopic surgery reduced postoperative pain and improved the surgical condition compared to conventional moderate neuromuscular blockade. However, the effect of neuromuscular blockade on robot-assisted thyroid surgery has not been studied yet.

There was concern about delayed recovery of muscle relaxation and respiratory failure due to deep neuromuscular blockade. However, the development of sugammadex (Bridion, Merck Sharp and Dohme - MSD, Oss, Netherlands) eliminated these concerns. Sugammadex dramatically reduced the recovery time from deep neuromuscular blockade.

ELIGIBILITY:
Inclusion Criteria:

* A. 20-70 yrs old patients scheduled for robot-assisted transaxillary thyroidectomy
* B. ASA(American Society of Anesthesiologists) classification: Ⅰ-Ⅲ
* C. Patients who voluntarily agree to participate in this clinical study.

Exclusion Criteria:

* A. Patients scheduled for radical neck node dissection
* B. Patients scheduled for co-operation of other organs or Patients with other accompanying cancers
* C. Patients with BMI(Body Mass Index) > 30 kg/m2
* D. Patients with history of Liver failure, Renal failure
* E. Patients who already have pain or paresthesia on chest, axilla, or neck.
* F. Patients with history of allergy to rocuronium or sugammadex
* G. Patients who cannot read the consent form (examples: Illiterate, foreigner)
* H. Pregnant woman, Lactating woman

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Postoperative pain: NRS | POD 1day
  Postoperative pain on POD 1day and POD 3days
  * assessed by Numeric Rating Scale (NRS)
  * score = 0~10 (No pain = 0, the worst pain = 10)
Postoperative pain: NRS | POD 3days
  Postoperative pain on POD 1day and POD 3days
  * assessed by Numeric Rating Scale (NRS)
  * score = 0~10 (No pain = 0, the worst pain = 10)

SECONDARY OUTCOMES:
Postoperative pain: NRS | 10 minutes after entering PACU(Post-Anesthetic Care Unit)
  * assessed by Numeric Rating Scale (NRS)
  * score = 0~10 (No pain = 0, the worst pain = 10)
Postoperative pain: NRS | POD 3months
  * assessed by Numeric Rating Scale (NRS)
  * score = 0~10 (No pain = 0, the worst pain = 10)
Postoperative sensory change | POD 1day
  Assessed by questionnaire. The questionnaire will ask the patients about the following items.
  1. the presence of abnormal sensation -> YES or NO
  2. characteristics of abnormal sensation -> 1. Numb 2. Tingling 3. Burning 4. Electricity 5. Other
  3. degree of abnormal sensation-> Scoring: 0~7 (No abnormal sensation = 0 . Very severe = 7)
Postoperative sensory change | POD 1day
  Assessed by pinprick test. The investigators will check the presence of postoperative sensory change through the pinprick test.-> Site: (1) Chest (2) Neck
Postoperative sensory change | POD 3days
  Assessed by questionnaire. The questionnaire will ask the patients about the following items.
  1. the presence of abnormal sensation -> YES or NO
  2. characteristics of abnormal sensation -> 1. Numb 2. Tingling 3. Burning 4. Electricity 5. Other
  3. degree of abnormal sensation-> Scoring: 0~7 (No abnormal sensation = 0 . Very severe = 7)
Postoperative sensory change | POD 3days
  Assessed by pinprick test. The investigators will check the presence of postoperative sensory change through the pinprick test.-> Site: (1) Chest (2) Neck
Postoperative sensory change | POD 3months
  Assessed by questionnaire. The questionnaire will ask the patients about the following items.
  1. the presence of abnormal sensation -> YES or NO
  2. characteristics of abnormal sensation -> 1. Numb 2. Tingling 3. Burning 4. Electricity 5. Other
  3. degree of abnormal sensation-> Scoring: 0~7 (No abnormal sensation = 0 . Very severe = 7)
Postoperative sensory change | POD 3months
  Assessed by pinprick test. The investigators will check the presence of postoperative sensory change through the pinprick test.-> Site: (1) Chest (2) Neck
Nausea/Vomiting | 10 minutes after entering PACU(Post-Anesthetic Care Unit)
  * Assessed by nausea/vomiting score
  * Score = 0~3
  * 0: no nausea
  * 1: mild nausea (no medication)
  * 2: severe nausea (anti-emetic used)
  * 3: retching and/or vomiting
Nausea/Vomiting | POD 1day
  * Assessed by nausea/vomiting score
  * Score = 0~3
  * 0: no nausea
  * 1: mild nausea (no medication)
  * 2: severe nausea (anti-emetic used)
  * 3: retching and/or vomiting
Nausea/Vomiting | POD 3days
  * Assessed by nausea/vomiting score
  * Score = 0~3
  * 0: no nausea
  * 1: mild nausea (no medication)
  * 2: severe nausea (anti-emetic used)
  * 3: retching and/or vomiting
The time from sugammadex injection to TOF ratio 0.9. | immediate postoperative
Number of patients with complications due to deep neuromuscular blockade (e.g. Respiratory failure, Desaturation) | From surgery to POD 3months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee J, Chung WY. Robotic thyroidectomy and neck dissection: past, present, and future. Cancer J. 2013 Mar-Apr;19(2):151-61. doi: 10.1097/PPO.0b013e31828aab61. PMID 23528724
- [Background] Lee J, Nah KY, Kim RM, Ahn YH, Soh EY, Chung WY. Differences in postoperative outcomes, function, and cosmesis: open versus robotic thyroidectomy. Surg Endosc. 2010 Dec;24(12):3186-94. doi: 10.1007/s00464-010-1113-z. Epub 2010 May 19. PMID 20490558
- [Background] Tae K, Ji YB, Cho SH, Lee SH, Kim DS, Kim TW. Early surgical outcomes of robotic thyroidectomy by a gasless unilateral axillo-breast or axillary approach for papillary thyroid carcinoma: 2 years' experience. Head Neck. 2012 May;34(5):617-25. doi: 10.1002/hed.21782. Epub 2011 Jun 17. PMID 21688343
- [Background] Kang SW, Jeong JJ, Nam KH, Chang HS, Chung WY, Park CS. Robot-assisted endoscopic thyroidectomy for thyroid malignancies using a gasless transaxillary approach. J Am Coll Surg. 2009 Aug;209(2):e1-7. doi: 10.1016/j.jamcollsurg.2009.05.003. Epub 2009 Jun 12. No abstract available. PMID 19632588
- [Background] Kim MH, Lee KY, Lee KY, Min BS, Yoo YC. Maintaining Optimal Surgical Conditions With Low Insufflation Pressures is Possible With Deep Neuromuscular Blockade During Laparoscopic Colorectal Surgery: A Prospective, Randomized, Double-Blind, Parallel-Group Clinical Trial. Medicine (Baltimore). 2016 Mar;95(9):e2920. doi: 10.1097/MD.0000000000002920. PMID 26945393
- [Background] Martini CH, Boon M, Bevers RF, Aarts LP, Dahan A. Evaluation of surgical conditions during laparoscopic surgery in patients with moderate vs deep neuromuscular block. Br J Anaesth. 2014 Mar;112(3):498-505. doi: 10.1093/bja/aet377. Epub 2013 Nov 15. PMID 24240315
- [Background] Dubois PE, Putz L, Jamart J, Marotta ML, Gourdin M, Donnez O. Deep neuromuscular block improves surgical conditions during laparoscopic hysterectomy: a randomised controlled trial. Eur J Anaesthesiol. 2014 Aug;31(8):430-6. doi: 10.1097/EJA.0000000000000094. PMID 24809482
- [Background] Jones RK, Caldwell JE, Brull SJ, Soto RG. Reversal of profound rocuronium-induced blockade with sugammadex: a randomized comparison with neostigmine. Anesthesiology. 2008 Nov;109(5):816-24. doi: 10.1097/ALN.0b013e31818a3fee. PMID 18946293
- [Background] Geldner G, Niskanen M, Laurila P, Mizikov V, Hubler M, Beck G, Rietbergen H, Nicolayenko E. A randomised controlled trial comparing sugammadex and neostigmine at different depths of neuromuscular blockade in patients undergoing laparoscopic surgery. Anaesthesia. 2012 Sep;67(9):991-8. doi: 10.1111/j.1365-2044.2012.07197.x. Epub 2012 Jun 14. PMID 22698066
- [Background] Welliver M, McDonough J, Kalynych N, Redfern R. Discovery, development, and clinical application of sugammadex sodium, a selective relaxant binding agent. Drug Des Devel Ther. 2009 Feb 6;2:49-59. doi: 10.2147/dddt.s2757. PMID 19920893